CLINICAL TRIAL: NCT07048171
Title: TO DETERMINE THE EFFECT OF ALLOGRAFT AND iPRF WITH OR WITHOUT COLLAGEN MEMBRANE ON HEALING OF APICOMARGINAL DEFECTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mareesha
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Apicomarginal Defects

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with apicomarginal defects receiving bone graft and iPRF with collagen membrane (Experimental): surgery performed using DFDBA bone graft and iPRF with collagen membrane
  Interventions: Procedure: Endodontic Micro-Surgery
- patients with apicomarginal defects receiving bone graft and iPRF without collagen membrane (Active Comparator): surgery performed using DFDBA bone graft and iPRF without collagen membrane
  Interventions: Procedure: Endodontic Micro-Surgery

INTERVENTIONS:
Procedure: Endodontic Micro-Surgery — Surgery performed using bone graft(DFDBA) and iPRF with collagen membrane in test group and bone graft and iPRF without collagen membrane in control group

SUMMARY:
To determine the effect of allograft and iPRF with or without collagen membrane on healing of apicomarginal defects : A Randomized Controlled Trial

DETAILED DESCRIPTION:
RATIONALE: - Apicomarginal defects are characterized by localized alveolar bone loss spanning the entire length of the root from the crestal alveolar bone to the apex of the tooth. These defects often present as a challenge in endodontic and periodontal therapy due to their extensive involvement of both the root apex and the periodontal tissues. .The use of guided tissue regeneration techniques has been proposed as an adjunct to endodontic surgery in order to promote bone healing Guided tissue regeneration (GTR) is a technique which prevent epithelial down growth, if the epithelial cells are excluded from a wound long enough for other cells types with regenerative potential to become established. Till date about 14 studies have been done on apicomarginal defects involving 12 on human and 2 on animal studies. Many studies have used either membrane alone , membrane and bone graft , only membrane or periosteal bone graft/ autologus platelet concentrate for promoting healing in such defects. .Both membrane ,graft as well as combination of membrane and graft may act a space maintainer to prevent epithelial migration .No study so far has compared three dimensional healing after endodontic surgery with adjunct use of graft with or without use of membrane in apicomarginal defects. Nevertheless there has been no study with the use of allograft and iPRF with collagen membrane versus allograft and iPRF in the healing of apicomarginal defects and quality of life assessment.

AIM To assess whether the application of allograft and iPRF with collagen membrane leads to improved healing outcomes and enhanced quality of life compared to the use of only allogafts and iPRF in patients of apicomarginal defects .

PRIMARY OBJECTIVE To evaluate the impact of application of allograft and iPRF with collagen membrane on buccal bone regeneration and 2d healing and 3d healing outcome using Rud and Molven et al. (1987). & modified PENN 3D criteria.

SECONDARY OBJECTIVE To compare quality of life of patients after periapical surgery with use of allograft and iPRF with collagen membrane and allograft and iPRF without collagen membrane in cases of apicomarginal defects .

SETTING: -Study will be conducted in Post Graduate Institute of Dental Sciences, Rohtak in the department of Conservative Dentistry & Endodontics.

STUDY DESIGN: - A randomized controlled trial

TIME FRAME: - 12Months

ELIGIBILITY:
Inclusion Criteria:

1. Patients with no general medical contraindications for oral surgical procedures (ASA-I and ASA-II according to the classification of the American Society of Anesthesiologist's).
2. Patients aged 18 years and above, presenting with chronic suppurative apical periodontitis in at least one tooth,
3. Radiographic evidence of apical radiolucency with periodontal pocket depth exceeding 6 mm confined to buccal aspect of the root.
4. Repeated abscess discharge despite satisfactory root canal treatment. 5.Patients with apicomarginal defects showing a denuded buccal bone plate

6.Failed primary root canal treatment 7.Adequate final restoration with no clinical evidence of coronal leakage.

Exclusion Criteria:

1. Clinical or radiographic evidence of root fracture.
2. Resorptive processes involving more than apical third of the root.
3. Chronic generalized periodontitis.
4. Failed previous endodontic surgery or failed root canal re-treatment.
5. Any systemic disease contraindicating oral surgery including uncontrolled diabetes and pregnancy, any condition effecting rate of healing like smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
Periapical healing assessment | Base line to 12 months
  Periapical healing comparison in 2 groups with buccal bone regeneration and 2d healing and 3d healing outcome using Rud and Molven et al. (1987). & modified PENN 3D criteria .

SECONDARY OUTCOMES:
Quality of life assessment | Base line to 12 months
  to assess pain, swelling, mouth opening and effect on daily activities of patient among test and control group using OHIP-14 questionnaire. Pain Assesment with Value 0 indicate no pain & 100 indicate maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India